CLINICAL TRIAL: NCT05578170
Title: Efficacy and Safety of Neoadjuvant Pembrolizumab in III-IVA Resectable Oral Squamous Cell Carcinoma
Acronym: PROBES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Liu xiqiang，MD, Doctor of Medicine，Chief Physician, Nanfang Hospital, Southern Medical University
Other Study IDs: NFEC-2022-082
Record Dates: First submitted 2022-10-08; First posted 2022-10-13 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Oral Cavity Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pembro Neoadjuvant + SOC Adjuvant
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Participants receive 200 mg pembrolizumab as a neoadjuvant by intravenous (IV) infusion administered on Day 1 of a 21-day cycle for 2 cycles before surgery.

SUMMARY:
The purpose of this prospective, single-center, single-arm, open-label II phase observation clinical trial is to evaluate the efficacy and safety of Pembrolizumab immunoadjuvant therapy in patients with stage III-IVA oral squamous cell carcinoma. The primary end point is the pathological tumor remission rate of the primary tumor and regional lymph nodes after neoadjuvant immunotherapy (pTR-2: the proportion of necrotic tumor cells, keratin fragments and giant cells in tissue sections > 50%). The secondary endpoints are 1-year disease-free survival (DFS), 1-year overall survival (OS) and the incidence of adverse events, compared with historical data. In addition, we will check the relevant immune indicators, such as PD-L1 and CPS scores.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Male and female
* Patients histologically or cytologically difined as oral cavity squamous cell carcinoma
* According to the American Joint Committee on Cancer ( AJCC 8th Edition ) , patients with resectable stage III-IVA OCSCC
* ECOG performance status ≤ 1
* Patients with normal bone marrow and organ function as defined below:

Blood routine examination:

1. Absolute neutrophil count ≥ 1.5×109/L;
2. Platelets ≥ 100.0×109/L;
3. Hemoglobin ≥ 9.0 g/dL.

Liver function:

1. Totle bilirubin ≤ 2.0×ULN(Upper Limit Of Normal);
2. Alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase

   * 2.5×ULN;
3. Albumin ≥ 2.8g/dL.

Renal function:

(1)Creatinine clearance rate > 60.0ml/min.

Coagulation function:

(1)International Normalized Ratio ≤ 1.5；Activated Partial Thromboplastin Time ≤ 1.5×ULN

* Prior to and during study, and lasting 120 days for the final utilization of pembrolizumab, patients approve of contraception
* Patients voluntarily agree to participate in the study and sign the informed consent form

Exclusion Criteria:

* Prior treatment for OCSCC (sugery, immunotherapy, radiotherapy, chemotherapy)
* Patients with metastatic OCSCC with an unknown primary tumor site
* Patients with infectious disease: AIDS, hepatitis, active tuberculosis
* Received a live vaccine within 30 days prior to the first dose of pembrolizumab. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, Bacillus Calmette-Guérin ( BCG ), typhoid vaccine, or attenuated flu vaccine
* 5.Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of pembrolizumab
* Currently receiving any other investigational agents
* Has a history of allergic reactions attributed to compounds of similar chemical of biologic composition to pembrolizumab or other agents used in the study
* Patients with ongoing or active infectoin requiring systemic therapy, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, underlying pulmonary disease, or psychiatric illness/social situations that would limit compliance with study requirements
* Has a or more active autoimmune disease
* Has a history( non-infectious ) pneumonitis that required steroids or current pneumonitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage III-IVA oral squamous cell carcinoma.(See Eligibility Criteria)
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of pathologic tumor response-2（pTR-2） | Up to 30 days post-sugery
  The proportion of participants with a pathologic tumor response-2（pTR-2）as assessed by the Central Pathologist at the time of definitive surgery. pTR-2 is defined as the proportion of necrotic tumor cells, keratin fragments and giant cells in tissue sections > 50%

SECONDARY OUTCOMES:
Disease-free Survival (DFS) | Up to 1 year
  DFS is the time from the date of randomization to the date of first record of any of the following events: disease progression; local or distant recurrence as assessed with imaging or biopsy as indicated; or death due to any cause
Overall Survival (OS) | Up to 1 year
  OS is the time from surgery to death due to any cause.
Adverse Events (AEs) | From time of first dose of study treatment until the end of follow-up (up to 1 year)
  Participants experiencing any sign, symptom, disease, or worsening of preexisting condition temporally associated with study therapy and irrespective of causality to study therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Liuxiqiang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No